CLINICAL TRIAL: NCT00270270
Title: A Double-Blind, Placebo-Controlled Study With Open-Label Follow-up to Determine the Safety and Efficacy of r-HuEPO in AIDS Patients With Anemia Induced by Their Disease and AZT Therapy
Brief Title: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa Versus Placebo for the Treatment of Anemia in AIDS (Acquired Immunodeficiency Syndrome) Patients With Anemia Caused by the Disease and by Zidovudine (AZT) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006070; NCT00547313 (obsolete NCT alias)
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Acquired Immunodeficiency Syndrome; Anemia
Keywords: erythropoietin; Anemia; Quality of Life; epoetin alfa; HIV; Zidovudine; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of epoetin alfa versus placebo in AIDS patients for the treatment of anemia that is a result of the disease or a result of zidovudine (AZT) treatment for AIDS. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
It is estimated that approximately 75% to 80% of patients with AIDS experience anemia, which can be caused by AIDS or by the therapy patients receive for AIDS treatment (for example, zidovudine [AZT]). Anemia is a condition in which a patient has below normal levels of hemoglobin, the substance in red blood cells that carries oxygen to all parts of the body. People with severe anemia may experience fatigue and shortness of breath with activity. Therefore, this condition can have a negative influence on a person's quality of life. Epoetin alfa, used to treat anemia, is a genetically engineered form of a natural hormone, erythropoietin, that stimulates red blood cell production. This is a randomized, double-blind, placebo-controlled study with an open-label follow-up period that is designed to evaluate the safety and effectiveness of epoetin alfa treatment compared with placebo treatment in patients with AIDS who are being treated with AZT. The study consists of three periods: a screening period to determine if patients are eligible for the study, a double-blind period, and an open-label period. During the double-blind period, patients are randomly assigned to one of two groups and receive either epoetin alfa (100 units per kilogram) or placebo injected into a vein (intravenously) three times per week for 12 weeks or until their hematocrit reaches 38% to 40%. In the open-label period, all patients receive epoetin alfa injected under the skin (subcutaneously) for up to 6 months at the dose needed to maintain hematocrit levels of 38% to 40%. Effectiveness will be determined by the change in hemoglobin, hematocrit, and reticulocyte count (laboratory tests used to evaluate the severity of anemia), transfusion requirements, and the patient's quality of life assessment. Safety assessments include the incidence and severity of adverse events during the study, results of clinical laboratory tests (hematology, biochemistry, and urinalysis), measurements of vital signs, electrocardiograms (ECGs) and physical examination findings. The study hypothesis is that for treatment of anemia in patients with AIDS who are receiving AZT therapy, epoetin alfa is superior to placebo, as measured by changes in hemoglobin, hematocrit, and reticulocyte count, transfusion requirements, and the patient's quality of life.

Double-blind period: epoetin alfa (100 units per kilogram [U/kg] of body weight) or placebo, injected intravenously three times a week for 12 weeks. Open-label period: epoetin alfa injected under the skin for up to 6 months, with dose adjustments in the range of 0 to 1,500 U/kg as needed to maintain hematocrit levels of 38% to 40%.

ELIGIBILITY:
Inclusion Criteria: - Patients with a confirmed diagnosis of AIDS, with a hematocrit <=30% - preferably dependent on transfusions - having a history of at least a 15% decrease in hematocrit since the beginning of AZT therapy, or have become dependent on transfusions - who are clinically stable for at least 1 month before study entry - females must be at least 1 year post-menopausal, surgically sterile, or practicing an effective method of birth control, and have a negative pregnancy test before study entry.

Exclusion Criteria: - Patients with a history of any primary blood disease - having any clinically significant disease or malfunction of the lungs, heart, hormones, neurological, gastrointestinal, reproductive or urinary systems, which is not caused by the AIDS infection - having uncontrolled high blood pressure - having anemia caused by conditions other than AIDS (for example, vitamin deficiency or bleeding from the gastrointestinal tract) - having a serum ferritin value <30 ng/mL or an iron/total iron-binding capacity (Fe/TIBC) ratio less than 15%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Study Completion 1989-07 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin, hematocrit, and reticulocyte count (laboratory tests used to evaluate the severity of anemia); Transfusion requirements; Safety evaluations including adverse events

SECONDARY OUTCOMES:
Patient's quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Ortho Biotech Products, L.P. Clinical Trial, Study Director — Ortho Biotech, Inc.

REFERENCES:
- See also: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa in Patients with Acquired Immune Deficiency Syndrome (AIDS) Who Are Receiving AZT Therapy (DB Phase) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=708&filename=CR006070_CSR.pdf
- See also: A Study to Evaluate the Safety and Efficacy of Epoetin Alfa in Patients with Acquired Immune Deficiency Syndrome (AIDS) Who Are Receiving AZT Therapy (DB Phase) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=708&filename=CR006070_CSR1.pdf